CLINICAL TRIAL: NCT00451204
Title: A Combination Trial of Copaxone Plus Estriol in RRMS
Brief Title: A Combination Trial of Copaxone Plus Estriol in Relapsing Remitting Multiple Sclerosis (RRMS)
Acronym: Estriol-MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Washington University School of Medicine (Other); University of Texas Southwestern Medical Center (Other); Ohio State University (Other); University of Medicine and Dentistry of New Jersey (Other); University of Chicago (Other); University of Utah (Other); Johns Hopkins University (Other); University of Kansas Medical Center (Other); University of Minnesota (Other); Mayo Clinic (Other); University of Colorado, Denver (Other); University of New Mexico (Other); University of Pennsylvania (Other); Dartmouth-Hitchcock Medical Center (Other); National Multiple Sclerosis Society (Other); National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Rhonda Voskuhl, Professor, Department of Neurology; Director Multiple Sclerosis Program, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NS051591 (NIH); R01NS051591 (NIH); RG3915 (Other Grant/Funding Number: NMSS)
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Results first posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; estrogen; estriol; progesterone
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Estriol; Estrogens; Sugars; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Estriol plus Copaxone injections QD (Active Comparator): Estriol Capsules (daily) plus Copaxone injections (daily). Progestin capsules given for 2 weeks every 3 months to avoid unopposed estrogens.
  Interventions: Drug: Estriol; Drug: Copaxone
- Placebo plus Copaxone injections QD (Placebo Comparator): Placebo Capsules (daily) plus Copaxone injections (daily). A second placebo capsule given for 2 weeks every 3 months.
  Interventions: Drug: Placebo; Drug: Copaxone

INTERVENTIONS:
Drug: Estriol — Estriol 8 mg capsule, once per day, duration of treatment is 2 years
  Other Names: E3; estrogen
  Arms: Estriol plus Copaxone injections QD
Drug: Placebo — Placebo capsule, once a day, treatment duration is 2 years
  Other Names: "sugar pill"
  Arms: Placebo plus Copaxone injections QD
Drug: Copaxone — Injection, once a day, all subjects
  Other Names: glatiramer acetate

SUMMARY:
This is a double-blinded, placebo controlled study of estriol pills versus placebo pills in relapsing remitting multiple sclerosis. The study treatment will be an added on to Copaxone injections in all subjects. The primary outcome measure is a reduction in relapses.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) relapses are known to be significantly decreased during pregnancy. This proposal will establish whether oral treatment with estriol, the major estrogen of pregnancy, induces a decrease in relapses in relapsing remitting multiple sclerosis (RRMS) subjects when used in combination with injectable Copaxone. Previously, in a pilot study, it has been demonstrated that treatment of RRMS subjects with oral estriol for six months resulted in a significant reduction in gadolinium enhancing lesions on serial brain MRIs (Annals of Neurology, 2002; 52:421-428) and caused a favorable shift in immune responses (Journal of Immunology, 2003; 171:6267-6274). This is an add-on study aiming to extend these previous findings by treating longer and focusing on clinical outcomes. The combination of Copaxone injection plus estriol pill (8 mg per day) will be compared to Copaxone injection plus placebo pill in a double blind trial. The duration of treatment will be two years and the primary outcome measure will be relapse rate. Other outcomes will include disability measures and brain MRI outcomes. Safety measures (blood tests and gynecologic evaluations) will also be followed and correlations will be made between serum estriol levels with efficacy and safety. The overall goal of this study will be the development of a new oral treatment, estriol, for RRMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remitting multiple sclerosis
* At least one relapse in the last two years

Exclusion Criteria:

* Patients treated in the past with total lymphoid irradiation, monoclonal antibody, T cell vaccination, cladribine, bone marrow transplantation, azathioprine, cyclophosphamide, methotrexate, mitoxantrone, cyclosporin or Tysabri
* Clinically significant diseases other than multiple sclerosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2007-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Voskuhl, M.D., Study Director — University of California, Los Angeles (UCLA), Los Angeles, CA; Anne Cross, M.D., Principal Investigator — Washington University, Saint Louis, MO; Elliot Frohman, M.D., Principal Investigator — University of Texas, Southwestern, Dallas, TX; Suhayl Dhib-Jalbut, M.D., Principal Investigator — Robert Wood Johnson Medical School, UMDNJ, New Brunswick, NJ; Michael Racke, M.D., Principal Investigator — Ohio State University; Anthony Reder, M.D., Principal Investigator — University of Chicago; John Rose, M.D., Principal Investigator — Western Institute for Biomedical Research, Salt Lake City, UT; Barbara Giesser, M.D., Principal Investigator — University of California, Los Angeles (UCLA), Los Angeles, CA; John Ratchford, M.D., Principal Investigator — Johns Hopkins, Baltimore, MD; Sharon Lynch, M.D., Principal Investigator — University of Kansas; Gareth Parry, M.D., Principal Investigator — University of Minnesota; Dean Wingerchuk, M.D., Principal Investigator — Mayo Clinic; John Corboy, M.D., Principal Investigator — University of Colorado, Denver; Corey Ford, M.D., Principal Investigator — University of New Mexico, Albuquerque; Dina Jacobs, M.D., Principal Investigator — University of Pennsylvania; Lloyd Kasper, M.D., Principal Investigator — Dartmouth University, Lebanon, NH
Locations (16):
- United States (15):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Dartmouth Medical School, Lebanon, New Hampshire
  - UMDNJ-Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Western Institute for Biomedical Research, Salt Lake City, Utah
- Montreal Neurological Institute, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Yes
Investigators interested in further research using the data should contact Dr. Voskuhl with proposed plans and request.

REFERENCES:
- [Background] Sicotte NL, Liva SM, Klutch R, Pfeiffer P, Bouvier S, Odesa S, Wu TC, Voskuhl RR. Treatment of multiple sclerosis with the pregnancy hormone estriol. Ann Neurol. 2002 Oct;52(4):421-8. doi: 10.1002/ana.10301. PMID 12325070
- [Background] Soldan SS, Alvarez Retuerto AI, Sicotte NL, Voskuhl RR. Immune modulation in multiple sclerosis patients treated with the pregnancy hormone estriol. J Immunol. 2003 Dec 1;171(11):6267-74. doi: 10.4049/jimmunol.171.11.6267. PMID 14634144
- [Background] Morales LB, Loo KK, Liu HB, Peterson C, Tiwari-Woodruff S, Voskuhl RR. Treatment with an estrogen receptor alpha ligand is neuroprotective in experimental autoimmune encephalomyelitis. J Neurosci. 2006 Jun 21;26(25):6823-33. doi: 10.1523/JNEUROSCI.0453-06.2006. PMID 16793889
- [Background] Tiwari-Woodruff S, Morales LB, Lee R, Voskuhl RR. Differential neuroprotective and antiinflammatory effects of estrogen receptor (ER)alpha and ERbeta ligand treatment. Proc Natl Acad Sci U S A. 2007 Sep 11;104(37):14813-8. doi: 10.1073/pnas.0703783104. Epub 2007 Sep 4. PMID 17785421
- [Background] Sicotte NL, Giesser BS, Tandon V, Klutch R, Steiner B, Drain AE, Shattuck DW, Hull L, Wang HJ, Elashoff RM, Swerdloff RS, Voskuhl RR. Testosterone treatment in multiple sclerosis: a pilot study. Arch Neurol. 2007 May;64(5):683-8. doi: 10.1001/archneur.64.5.683. PMID 17502467
- [Background] Gold SM, Sasidhar MV, Morales LB, Du S, Sicotte NL, Tiwari-Woodruff SK, Voskuhl RR. Estrogen treatment decreases matrix metalloproteinase (MMP)-9 in autoimmune demyelinating disease through estrogen receptor alpha (ERalpha). Lab Invest. 2009 Oct;89(10):1076-83. doi: 10.1038/labinvest.2009.79. Epub 2009 Aug 10. PMID 19668239
- [Background] Ziehn MO, Avedisian AA, Dervin SM, O'Dell TJ, Voskuhl RR. Estriol preserves synaptic transmission in the hippocampus during autoimmune demyelinating disease. Lab Invest. 2012 Aug;92(8):1234-45. doi: 10.1038/labinvest.2012.76. Epub 2012 Apr 23. PMID 22525427
- [Background] Spence RD, Hamby ME, Umeda E, Itoh N, Du S, Wisdom AJ, Cao Y, Bondar G, Lam J, Ao Y, Sandoval F, Suriany S, Sofroniew MV, Voskuhl RR. Neuroprotection mediated through estrogen receptor-alpha in astrocytes. Proc Natl Acad Sci U S A. 2011 May 24;108(21):8867-72. doi: 10.1073/pnas.1103833108. Epub 2011 May 9. PMID 21555578
- [Result] Voskuhl RR, Wang H, Wu TC, Sicotte NL, Nakamura K, Kurth F, Itoh N, Bardens J, Bernard JT, Corboy JR, Cross AH, Dhib-Jalbut S, Ford CC, Frohman EM, Giesser B, Jacobs D, Kasper LH, Lynch S, Parry G, Racke MK, Reder AT, Rose J, Wingerchuk DM, MacKenzie-Graham AJ, Arnold DL, Tseng CH, Elashoff R. Estriol combined with glatiramer acetate for women with relapsing-remitting multiple sclerosis: a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Jan;15(1):35-46. doi: 10.1016/S1474-4422(15)00322-1. Epub 2015 Nov 29. PMID 26621682

RESULTS

PARTICIPANT FLOW:
Groups:
- Estriol Capsules Plus Copaxone Injections: Estriol: Estriol 8 mg capsule, once per day, duration of treatment is 2 years
- Placebo Capsules Plus Copaxone Injections: Placebo: Placebo capsule, once per day, treatment duration is 2 years
Period: Overall Study
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Started | 82 | 76
Completed | 60 (60 completed the study but 3 stopped study drug(s) early) | 56
Not Completed | 22 | 20
Not completed — Adverse Event | 4 | 6
Not completed — Lack of Efficacy | 4 | 4
Not completed — Lost to Follow-up | 4 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Patient refusal | 8 | 4
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Relapsing remitting multiple sclerosis women aged 18 to 50 years.
Groups:
- Placebo Capsules Plus Copaxone Injections: Placebo: Placebo capsule, once a day, treatment duration is 2 years
- Total: Total of all reporting groups
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections | Total
Number analyzed (Participants) | 82 | 76 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 76 | 158
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (7.6) | 37.1 (7.3) | 37.4 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 76 | 158
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 82 | 76 | 158

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Relapse, Annualized Relapse Rate
Description: A confirmed relapse was defined as new neurological symptoms or worsening of pre-existing symptoms, lasting at least 48 hours in a subject who had been neurologically stable or improving in the previous 30 days, accompanied by objective change in the neurological examination (worsening of 0.5 points on the EDSS or worsening by 1.0 or more points on the pyramidal, cerebellar, brainstem or visual functional system scores), not due to fatigue alone and not associated with fever or infection.
Time Frame: 24 months
Population: Included all as intention to treat
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Number analyzed (Participants) | 82 | 76
relapses per year | 0.25 [0.17 to 0.37] | 0.37 [0.25 to 0.53]
Statistical Analysis 1: Comparison: Estriol Capsules Plus Copaxone Injections vs Placebo Capsules Plus Copaxone Injections; Test type: Superiority or Other; p = 0.077, negative binomial regression; adjusted for age, BL EDSS score, # of relapses in previous 12 mo, time since dx, previous glatiramer acetate tx, and previous interferon beta tx; Rate ratio = 0.63, 95% CI 2-sided [0.37 to 1.05]

2. Secondary Outcome: Relapse Event, Annualized Relapse Rate
Description: Met all criteria for relapse except not confirmed to have increase in EDSS by an independent examiner.
Time Frame: 24 months
Population: Included all as intention to treat.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Number analyzed (Participants) | 82 | 76
relapses per year | 0.32 [0.22 to 0.46] | 0.46 [0.32 to 0.65]
Statistical Analysis 1: Comparison: Estriol Capsules Plus Copaxone Injections vs Placebo Capsules Plus Copaxone Injections; Test type: Superiority or Other; p = 0.098, negative binomial regression; adjusted for age, BL EDSS score, # of relapses in previous 12 months, time since dx, previous GA treatment, and previous interferon beta treatment; Rate ratio = 0.65, 95% CI 2-sided [0.39 to 1.08]

3. Secondary Outcome: Confirmed Relapse, Probability of First Relapse
Time Frame: 24 months
Population: All included as intention to treat
Measure: Mean (95% Confidence Interval); unit: probability of relapse at 24 months
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Number analyzed (Participants) | 82 | 76
probability of relapse at 24 months | 33.3 [23.8 to 45.4] | 42.9 [32.1 to 55.5]
Statistical Analysis 1: Comparison: Estriol Capsules Plus Copaxone Injections vs Placebo Capsules Plus Copaxone Injections; Test type: Superiority or Other; p = 0.096, negative binomial regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.63, 95% CI 2-sided [0.36 to 1.09]

4. Secondary Outcome: Relapse Event, Probability of First Relapse Event
Time Frame: 24 months
Population: Included all as intention to treat
Measure: Mean (95% Confidence Interval); unit: probability of relapse event at 24 mo
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Number analyzed (Participants) | 82 | 76
probability of relapse event at 24 mo | 40.5 [30.0 to 53.0] | 46.9 [35.9 to 59.3]
Statistical Analysis 1: Comparison: Estriol Capsules Plus Copaxone Injections vs Placebo Capsules Plus Copaxone Injections; Test type: Superiority or Other; p = 0.179, negative binomial regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.70, 95% CI 2-sided [0.42 to 1.17]

5. Other Pre Specified Outcome: Confirmed Relapse, Annualized Relapse Rate
Description: as for outcome 1
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: relapses per year
Groups:
- Estriol Capsules Plus Copaxone Injections: Estriol 8 mg capsule, once per day, duration of treatment is 2 years
- Placebo Capsules Plus Copaxone Injections: Placebo capsule, once a day, treatment duration is 2 years
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Number analyzed (Participants) | 82 | 76
relapses per year | 0.25 [0.16 to 0.40] | 0.48 [0.33 to 0.69]
Statistical Analysis 1: Comparison: Estriol Capsules Plus Copaxone Injections vs Placebo Capsules Plus Copaxone Injections; Test type: Superiority or Other; p = 0.016, negative binomial regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.49, 95% CI 2-sided [0.28 to 0.88]

6. Other Pre Specified Outcome: Relapse Event, Annualized Relapse Rate
Description: Met all criteria for relapse except not confirmed to have increase in EDSS by an independent examiner.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Number analyzed (Participants) | 82 | 76
relapses per year | 0.33 [0.22 to 0.50] | 0.61 [0.44 to 0.84]
Statistical Analysis 1: Comparison: Estriol Capsules Plus Copaxone Injections vs Placebo Capsules Plus Copaxone Injections; Test type: Superiority or Other; p = 0.012, negative binomial regression; [statistical method as in outcome 2, analysis 1]; Rate ratio = 0.52, 95% CI 2-sided [0.31 to 0.86]

ADVERSE EVENTS:
Time Frame: After enrollment, during the 24-month treatment period
Description: An adverse event is any condition that occurs after enrollment, whether or not considered related to study treatment.
Arm/Group | Estriol Capsules Plus Copaxone Injections | Placebo Capsules Plus Copaxone Injections
Serious Adverse Events (participants affected / at risk) | 8/82 | 10/76
Other Adverse Events (participants affected / at risk) | 76/82 | 67/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estriol Capsules Plus Copaxone Injections (N=82) | Placebo Capsules Plus Copaxone Injections (N=76)
MS Relapse (hospitalization) (Nervous system disorders) | 2 (2) | 5 (6)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Migraine headache related eye pain (Eye disorders) | 1 (1) | 0 (0)
Heart Failure/ pace maker implantation (Cardiac disorders) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Accidentally took other's drug (Investigations) | 0 (0) | 1 (1)
Acute appendicitis (Infections and infestations) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
car accident related body numbness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Right Knee Replacemebt (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estriol Capsules Plus Copaxone Injections (N=82) | Placebo Capsules Plus Copaxone Injections (N=76)
Upper respiratory Infection (Infections and infestations) | 22 (33) | 26 (38)
GA injection area abnormalities (Skin and subcutaneous tissue disorders) | 21 (25) | 12 (15)
Irregular menses/ spotting (Reproductive system and breast disorders) | 19 (26) | 3 (4)
Urinary tract infection (Renal and urinary disorders) | 15 (23) | 10 (16)
Fatigue (General disorders) | 13 (15) | 8 (10)
Depression/ Anxiety (Psychiatric disorders) | 12 (14) | 9 (10)
Menstrual flow amount increased (Reproductive system and breast disorders) | 11 (12) | 6 (8)
Headache (General disorders) | 9 (11) | 11 (12)
Nausea/ vomitting (Gastrointestinal disorders) | 7 (9) | 5 (5)
GA injection systemic reaction (SOB, hot flashes) (General disorders) | 7 (7) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (14)
Arm/ leg numbness, tingling (Nervous system disorders) | 6 (7) | 7 (10)
Gastroenteritis (Gastrointestinal disorders) | 5 (7) | 3 (4)
Dizziness (Nervous system disorders) | 4 (5) | 7 (10)
Vision problem (blurry, double) (Eye disorders) | 4 (6) | 7 (7)
Back Pain (General disorders) | 4 (5) | 5 (5)
Menstrual cramp (Reproductive system and breast disorders) | 4 (4) | 4 (5)
Insomnia (General disorders) | 4 (4) | 4 (4)
Heart palpitation (Cardiac disorders) | 2 (2) | 4 (4)
Shingles (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Vaginal infection (Reproductive system and breast disorders) | 1 (1) | 8 (9)
Uterus, endometrial thickness > 8mm (ultrasound) (Reproductive system and breast disorders) | 24 (29) | 27 (36)
Uterus, endometrial biopsies performed (Reproductive system and breast disorders) | 9 (11) | 6 (8)
Uterus, fibroibds (ultrasound) (Reproductive system and breast disorders) | 8 (10) | 8 (11)
Fibrocystic disease on clinical exam (Reproductive system and breast disorders) | 5 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No